CLINICAL TRIAL: NCT07392502
Title: Telerehabilitation for Shoulder Surgery Recovery: A Randomized Trial Assessing the Effectiveness of the Band Connect Platform
Brief Title: Telerehabilitation for Shoulder Surgery Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-01417
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (Active Comparator): Individuals in the control arm will complete standard physical therapy sessions.
  Interventions: Behavioral: Physical Therapy
- Band Connect Intervention (Experimental): Individuals in the experimental arm will complete standard physical therapy sessions while using the Band Connect device, which allows for direct measurement of patient force generated as well as positioning during the completion of physical therapy exercises.
  Interventions: Device: Band Connect; Behavioral: Physical Therapy

INTERVENTIONS:
Device: Band Connect — The Band Connect device has two main components: smart handles and resistance bands in varying lengths and resistance. The smart handles transfer data back to a phone app, which provides the patient instructions for their prescribed treatment as well as simulated biofeedback to ensure appropriate technique. The sensor function of Band Connect allows physical therapists to track participant movements to assess physical therapy activity. No video is being recorded of the participant.
  Arms: Band Connect Intervention
Behavioral: Physical Therapy — Standard physical therapy exercises for rotator cuff surgery rehabilitation.

SUMMARY:
This study aims to evaluate the effectiveness of a telerehabilitation protocol utilizing the Band Connect platform in patient recovery following rotator cuff repair surgery. This will be a randomized control trial with patients assigned into a traditional rehabilitation or a telerehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled for primary arthroscopic rotator cuff repair Surgery to be performed by Dr. Young Kwon, Dr. Mandeep Virk, Dr. Dennis DeBernardis, or Dr. Jie Yao
* Planning to complete postoperative physical therapy at selected NYU physical therapy locations
* Access to home internet and a wireless cell phone compatible with the Band Connect App

Exclusion Criteria:

* Patients undergoing revision RCR
* Patients whose post operative rehabilitation has to be delayed or modified.
* Pregnant individuals
* Shoulder injuries related to workers compensation or involved in any pending litigation
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in American Shoulder and Elbow Surgeons (ASES) | Baseline, Month 6
  The ASES is a 17-item questionnaire measuring shoulder pain and function. The total score is standardized into a 0-100 scale; higher scores indicate less pain/greater function.

SECONDARY OUTCOMES:
Change in Visual Analogue Scale (VAS) Pain Score | Baseline, Month 6
  Pain is rated on a scale from 0-100; higher scores indicate greater pain. Participants rate pain specific to the shoulder that was operated on.
Change in PROMIS Upper Extremity - Short Form 7a Score | Baseline, Month 6
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Upper Extremity - Short Form 7a comprises 7 questions assessing functionality of upper extremities. The raw score is standardized to a total score from 0-100 with a mean of 50 and standard deviation of 10. Higher scores indicate greater functionality of upper extremities.
Change in Days Per Week of Physical Therapy | Baseline, Month 6
  Number of days per week physical therapy exercises were completed at home.
Change in Intensity of Physical Therapy | Baseline, Month 6
  Participants rank the intensity on a scale from 0 (not intense) to 10 (intenst).

CONTACTS AND LOCATIONS:
Overall Officials: Young Kwon, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 3 months to 5 years after publication, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: young.kwon@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to young.kwon@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.